CLINICAL TRIAL: NCT01894828
Title: The Effect of Nutritional Supplementation in Cancer Patients With no Clinical Signs of Malnutrition
Brief Title: Nutritional Supplementation in Patients With no Signs of Malnutrition
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MedSource Polska (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Nutri01
Record Dates: First submitted 2013-07-04; First posted 2013-07-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Primary Neoplasm; Secondary Neoplasm; Abdominal Neoplasm
Keywords: Nutritional support; Gastrointestinal cancer; Malnutrition
MeSH Terms: conditions — Neoplasm Metastasis; Abdominal Neoplasms; Gastrointestinal Neoplasms; Malnutrition | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutritional supplements (Active Comparator): Patients are asked to drink two 200ml bottles of nutritional supplement daily
  Interventions: Dietary Supplement: Nutritional supplements
- Control (No Intervention): Patients are asked to keep on to their normal diet. No supplementation is introduced

INTERVENTIONS:
Dietary Supplement: Nutritional supplements — Patients are asked to drink two 200ml bottles of nutritional supplement daily for 14 days before surgery
  Arms: Nutritional supplements

SUMMARY:
The aim of the study was to assess the effect of nutritional supplementation on nutritional status and postoperational complications in cancer patients with no clinical signs of malnutrition

DETAILED DESCRIPTION:
In previous psychological studies our team found high level psychological stress in over 60% of cancer patients. This may cause numerous problems including anorexia, which together with biological disturbances can initiate cancer related catabolism even when it can not yet be seen. In this study we want to answer the question if oral nutritional supplementation can help the patient overcome the catabolism in its initial phase and improve nutritional status, which would result in reduced number of postoperational complications

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary resectable gastrointestinal and abdominal malignancy
* No signs of malnutrition at qualification for surgery
* General performance >70 Karnofsky scale
* Informed consent

Exclusion Criteria:

* history of radio or chemotherapy
* signs of mechanical ileus
* other major gastrointestinal diseases
* type 1 diabetes
* autoimmunological diseases requiring systemic steroids
* signs of infection
* renal and/or liver failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Improvement of nutritional status | After 14 days
  The aim of the study was to assess if nutritional supplementation improves nutritional status of patients with no clinical signs of malnutrition. Nutritional status improvement will be assessed by change in anthropometric (body weight (kg)) and laboratory (albumin, total protein, transferrin level, total lymphocyte count) parameters.

SECONDARY OUTCOMES:
Reducing number of complications | 30 days after surgery
  To assess if improvement of nutritional status is connected with reduced number of postoperative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Kabata, MD, Principal Investigator — Department of Surgical Oncology Medical University of Gdańsk; Tomasz Jastrzębski, Prof., Study Director — Department of Surgical Oncology Medical University of Gdańsk
Locations (1):
- Department of Surgical Oncology Medical University of Gdańsk, Gdansk, Pomeranian Voivodeship, Poland